CLINICAL TRIAL: NCT04487158
Title: Integrating Small Changes and Positive Psychology to Improve Treatment Readiness: A 12 Month Randomized Controlled Trial
Brief Title: Integrating Small Changes and Positive Psychology to Improve Treatment Readiness: A Weight Loss Trial
Acronym: INSPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lesley Lutes, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-02665
Record Dates: First submitted 2020-06-10; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: Behavioral Intervention; Psychological Intervention; Weight Management
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Changes (Active Comparator)
  Interventions: Behavioral: Small Changes
- INSPIRE (Experimental)
  Interventions: Behavioral: INSPIRE

INTERVENTIONS:
Behavioral: Small Changes — The Small Changes program is an evidence-based 6-month weight-management program. The program runs weekly for 3 months followed by by-weekly contact for 3-months (1x in-person group and 1x phone call). This program uses behaviour change strategies to help with weight loss. The Small Changes approach is different from traditional dieting programs because it encourages modest changes to diet and physical activity which are not overly taxing to maintain. Participants are asked to reduce their nutritional intake by 200-400 calories per day. You will also be asked to increase their daily step count by 2000-3000 steps. Weekly intervention topics include: Monitoring, Nutrition, Physical Activity, Breaking the Chain, External Cues, Mindful Eating, Body Image, Stress, Sleep, Social Support, Social Eating, and the Stoplight Guide.
  Arms: Small Changes
Behavioral: INSPIRE — The INSPIRE program is a modification to the Small Changes program. It combines elements of positive psychology and behaviour change to help with weight loss. The first four weeks of the program are oriented towards improving well-being and include topics such as values, self-compassion/mindfulness, character strengths, and gratitude. The remaining 8 weeks mirrors the Small Changes program in making modest changes to diet and physical activity to achieve weight loss. Participants are asked to reduce their nutritional intake by 200-400 calories per day. Participants will also be asked to increase their daily step count by 2000-3000 steps.
  Arms: INSPIRE

SUMMARY:
The study is designed to compare short- and long-term changes in body weight (kg) and subjective well-being in adult females with obesity who have been randomized to receive one of two 6-month treatment conditions: INSPIRE or Small Changes. The Small Changes approach is an evidence-based behavioural weight management program that uses relative and modest changes in nutrition and physical activity to produce a caloric deficit. The INSPIRE program is a modification of the Small Changes program that spends the first four weeks on improving well-being via psychological interventions.

DETAILED DESCRIPTION:
Rates of obesity continues to rise in Canada and worldwide, which is related to the presence and increased severity of multiple co-morbid illnesses as well as a reduction in overall quality and quantity of life. Traditional behavioural interventions have demonstrated efficacy in producing initial weight loss; however, a continued challenge for these programs is long-term weight loss maintenance. The Small Changes program is an alternative approach to weight loss that encourages modest changes to nutrition and physical activity that are sustainable long-term. Although promising, this approach has failed to consistently demonstrate clinically significant weight loss. It has been suggested that psychological factors, such as low levels of subjective well-being (negative affect, positive affect, and life satisfaction), may work in opposition of an individual's weight management goals. Thus, the integration of psychological interventions with a Small Changes approach has the potential to improve well-being and weight loss concurrently. Based on previous research, psychological interventions may be effectively utilized if they are implemented at the beginning of an intervention where early changes in well-being promote greater adherence to health behaviour change. To date, no behavioural intervention that integrates psychological approaches at treatment outset has been evaluated. The primary aim of the study is to determine the feasibility, acceptability, and efficacy of a novel group-based integrative behavioural and psychological intervention (INSPIRE) on change in weight and subjective well-being outcomes compared to an evidence-based behavioural intervention for weight loss (Small Changes).

ELIGIBILITY:
Inclusion Criteria:

* Female between the ages of 25 to 75
* BMI between 30 and 45
* Not currently participating in any other weight management programs
* Self-reports wanting to lose weight
* Willing to follow recommendations in the study protocol and attend weekly group intervention for 12 weeks and a 3-month follow-up group (one in-person group per month and one phone call per month)
* Ability to attend 4 assessment appointments over the course of the study period (at baseline, 3-months, 6-months, 12-months).
* Willing to be randomized into any of the two study arms and willing to adhere to guidelines and recommendations associated with the study arm they are randomized into

Exclusion Criteria:

* Cannot commit to weekly group times. Participants must be available for at least one group time of each intervention arm in order to be eligible to participate.
* Participated in a weight loss intervention in the past six months
* Participants who are pregnant (or less than 6 months post partum) or planning to become pregnant in the next 12 months
* Weight loss of > 5kg (~11 lb) in the previous 6 months
* History of, or current, clinically diagnosed eating disorder or exhibiting clinical symptoms of an eating disorder but undiagnosed (EDE-Q ≥ 4.0 unless clinical judgement indicates otherwise)
* Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (as measured by the PAR-Q+) where a doctor's note is not provided
* Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg
* If any of the following medical conditions are present: Insulin dependent diabetes; Previous surgical procedure for weight loss; Major surgery within the previous 6 months; A history of heart problems (e.g., angina, bypass surgery, myocardial infarction) within the previous 6 months; Implanted cardiac defibrillator or pacemaker; Currently (or within the past 5 years) being treated for cancer; Inflammatory Bowel Disease (i.e., chronic inflammatory gastrointestinal disease such as Crohn's Disease or Ulcerative Colitis); Chronic Pain (e.g., fibromyalgia) that would prevent the participant from engaging in physical activity
* The participant is currently experiencing elevated symptoms of depression
* The participant is planning to move within the study period
* The participant consumes more than 14 alcoholic drinks per week or more than 3 drinks per day

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as female
Enrollment: 60 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline weight (self-report) | 3 months
  (kg)
Change from baseline weight (self-report) | 6 months
  (kg)
Change from baseline weight | 9 months
  (kg)
Change from baseline weight | 12 months
  (kg)

SECONDARY OUTCOMES:
Change from Baseline on the Satisfaction with Life Scale | 3 months
  The Satisfaction with Life Scale is 5-item questionnaire used to assess life satisfaction which is a component of subjective well-being. Total scores range from 5 to 35 with higher scores indicating greater life satisfaction.
Change from Baseline on the Satisfaction with Life Scale | 6 months
  The Satisfaction with Life Scale is 5-item questionnaire used to assess life satisfaction which is a component of subjective well-being. Total scores range from 5 to 35 with higher scores indicating greater life satisfaction.
Change from Baseline on the Satisfaction with Life Scale | 12 months
  The Satisfaction with Life Scale is 5-item questionnaire used to assess life satisfaction which is a component of subjective well-being. Total scores range from 5 to 35 with higher scores indicating greater life satisfaction.
Change from Baseline on the Scale of Positive and Negative Experiences | 3 months
  The Scale of Positive and Negative Experiences 12-item self-report measure that will be used to measure two components of subjective well-being (positive affect and negative affect). The 12-items load onto two sub-scales: one pertaining to Positive Affect and the other pertaining to Negative Affect. Both subscales range from 6 to 30. Higher scores on these two sub-scales indicate greater experiences of either positive or negative affect states (i.e., higher scores on the SPANE-PA scale indicates greater frequency of experiencing positive emotions).
Change from Baseline on the Scale of Positive and Negative Experiences (SPANE) | 6 months
  The Scale of Positive and Negative Experiences is 12-item self-report measure that will be used to measure two components of subjective well-being (positive affect and negative affect). The 12-items load onto two sub-scales: one pertaining to Positive Affect and the other pertaining to Negative Affect. Both subscales range from 6 to 30. Higher scores on these two sub-scales indicate greater experiences of either positive or negative affect states (i.e., higher scores on the SPANE-PA scale indicates greater frequency of experiencing positive emotions).
Change from Baseline on the Scale of Positive and Negative Experiences (SPANE) | 12 months
  The Scale of Positive and Negative Experiences is 12-item self-report measure that will be used to measure two components of subjective well-being (positive affect and negative affect). The 12-items load onto two sub-scales: one pertaining to Positive Affect and the other pertaining to Negative Affect. Both subscales range from 6 to 30. Higher scores on these two sub-scales indicate greater experiences of either positive or negative affect states (i.e., higher scores on the SPANE-PA scale indicates greater frequency of experiencing positive emotions).

OTHER OUTCOMES:
Change from Baseline in Waist Circumference | 9 months
  (cm)
Change from Baseline in Waist Circumference | 12 months
  (cm)
Change from Baseline in Blood Pressure | 9 months
  Systolic and Diastolic Blood Pressure
Change from Baseline in Blood Pressure | 12 months
  Systolic and Diastolic Blood Pressure
Change from Baseline in Heart Rate | 9 months
Change from Baseline in Heart Rate | 12 months
Change from Baseline on the Self-Compassion Scale | 3 months
  The Self-Compassion Scale is a 26-item self-report measure which will be used to measure how an individual responds and acts towards themselves during difficult times. Total score ranges from 5 to 30 with higher scores indicating greater self-compassion.
Change from Baseline on the Self-Compassion Scale | 6 months
  The Self-Compassion Scale is a 26-item self-report measure which will be used to measure how an individual responds and acts towards themselves during difficult times. Total score ranges from 5 to 30 with higher scores indicating greater self-compassion.
Change from Baseline on the Self-Compassion Scale | 12 months
  The elf-Compassion Scale is a 26-item self-report measure which will be used to measure how an individual responds and acts towards themselves during difficult times. Total score ranges from 5 to 30 with higher scores indicating greater self-compassion.
Change from Baseline on the New General Self-Efficacy Scale | 3 months
  The New General Self-Efficacy is an 8-item self-report questionnaire that will be used to measure general self-efficacy. Total scores range from 8 to 40 with higher scores indicating greater general self-efficacy.
Change from Baseline on the New General Self-Efficacy Scale | 6 months
  The New General Self-Efficacy is an 8-item self-report questionnaire that will be used to measure general self-efficacy. Total scores range from 8 to 40 with higher scores indicating greater general self-efficacy.
Change from Baseline on the New General Self-Efficacy Scale | 12 months
  The New General Self-Efficacy is an 8-item self-report questionnaire that will be used to measure general self-efficacy. Total scores range from 8 to 40 with higher scores indicating greater general self-efficacy.
Change from Baseline on the Self-Efficacy for Exercise Scale | 3 months
  The Self-Efficacy for Exercise Scale is a 9-item self-report questionnaire that will be used to measure self-efficacy for exercise. Total scores range from 0 to 90 with higher scores representative of greater exercise-related self-efficacy.
Change from Baseline on the Self-Efficacy for Exercise Scale | 6 months
  The Self-Efficacy for Exercise Scale is a 9-item self-report questionnaire that will be used to measure self-efficacy for exercise. Total scores range from 0 to 90 with higher scores representative of greater exercise-related self-efficacy.
Change from Baseline on the Self-Efficacy for Exercise Scale | 12 months
  The Self-Efficacy for Exercise Scale is a 9-item self-report questionnaire that will be used to measure self-efficacy for exercise. Total scores range from 0 to 90 with higher scores representative of greater exercise-related self-efficacy.
Change from Baseline on the Weight Efficacy Lifestyle Questionnaire Short-Form | 3 months
  The Weight Efficacy Lifestyle Questionnaire Short-Form will be used to measure a specific form of self-efficacy related to eating habits. The WEL-SF is an 8-item measure with total scores ranging from 0 to 80 where higher scores are indicative of greater self-efficacy for eating habits.
Change from Baseline on the Weight Efficacy Lifestyle Questionnaire Short-Form | 6 months
  The Weight Efficacy Lifestyle Questionnaire Short-Form will be used to measure a specific form of self-efficacy related to eating habits. The WEL-SF is an 8-item measure with total scores ranging from 0 to 80 where higher scores are indicative of greater self-efficacy for eating habits.
Change from Baseline on the Weight Efficacy Lifestyle Questionnaire Short-Form | 12 months
  The Weight Efficacy Lifestyle Questionnaire Short-Form will be used to measure a specific form of self-efficacy related to eating habits. The WEL-SF is an 8-item measure with total scores ranging from 0 to 80 where higher scores are indicative of greater self-efficacy for eating habits.
Change from Baseline on the Three Factor Eating Questionnaire-Revised | 3 months
  The Three Factor Eating Questionnaire-Revised is an 18-item self-report measure of the cognitive and behavioural components of eating across three factors: Cognitive Restraint, Uncontrolled Eating, and Emotional Eating. Each subscale ranges from 1 to 4 (mean of all item on each subscale) with higher scores indicating greater endorsement of the subscale domain. Higher scores on the Cognitive Restraint represent greater cognitive restraint. Higher scores on the Uncontrolled subscale represent greater experiences with uncontrolled eating. Higher scores on the Emotional Eating subscale represent greater experiences with emotional eating.
Change from Baseline on the Three Factor Eating Questionnaire-Revised | 6 months
  The Three Factor Eating Questionnaire-Revised is an 18-item self-report measure of the cognitive and behavioural components of eating across three factors: Cognitive Restraint, Uncontrolled Eating, and Emotional Eating. Each subscale ranges from 1 to 4 (mean of all item on each subscale) with higher scores indicating greater endorsement of the subscale domain. Higher scores on the Cognitive Restraint represent greater cognitive restraint. Higher scores on the Uncontrolled subscale represent greater experiences with uncontrolled eating. Higher scores on the Emotional Eating subscale represent greater experiences with emotional eating.
Change from Baseline on the Three Factor Eating Questionnaire-Revised | 12 months
  The Three Factor Eating Questionnaire-Revised is an 18-item self-report measure of the cognitive and behavioural components of eating across three factors: Cognitive Restraint, Uncontrolled Eating, and Emotional Eating. Each subscale ranges from 1 to 4 (mean of all item on each subscale) with higher scores indicating greater endorsement of the subscale domain. Higher scores on the Cognitive Restraint represent greater cognitive restraint. Higher scores on the Uncontrolled subscale represent greater experiences with uncontrolled eating. Higher scores on the Emotional Eating subscale represent greater experiences with emotional eating.
Change from Baseline on the Food Cravings Inventory | 3 months
  The Food Cravings Inventory is a 33-item self-report measure of food cravings. Total score ranges from 33 to 165 with higher scores indicative of greater food cravings.
Change from Baseline on the Food Cravings Inventory | 6 months
  The Food Cravings Inventory is a 33-item self-report measure of food cravings. Total score ranges from 33 to 165 with higher scores indicative of greater food cravings.
Change from Baseline on the Food Cravings Inventory | 12 months
  The Food Cravings Inventory is a 33-item self-report measure of food cravings. Total score ranges from 33 to 165 with higher scores indicative of greater food cravings.
Change from Baseline on Objective Mean Step Count across 7 days | 3 months
  Step count from pedometers will be recorded daily and averaged across each week.
Change from Baseline on the Body Shape Questionnaire | 3 months
  The Body Shape Questionnaire is a 34-item self-report questionnaire of cognitively-based body dissatisfaction. Total scores range from 34 to 170 with higher scores indicative of greater body dissatisfaction.
Change from Baseline on the Body Shape Questionnaire | 6 months
  The Body Shape Questionnaire is a 34-item self-report questionnaire of cognitively-based body dissatisfaction. Total scores range from 34 to 170 with higher scores indicative of greater body dissatisfaction.
Change from Baseline on the Body Shape Questionnaire | 12 months
  The Body Shape Questionnaire is a 34-item self-report questionnaire of cognitively-based body dissatisfaction. Total scores range from 34 to 170 with higher scores indicative of greater body dissatisfaction.
Change from Baseline in Resting Metabolic Rate | 9 months
  Resting Metabolic Rate will be reported as kcal/day measured by indirect calorimetry
Change from Baseline in Resting Metabolic Rate | 12 months
  Resting Metabolic Rate will be reported as kcal/day measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Lutes, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No